CLINICAL TRIAL: NCT05195034
Title: Effect of Dexmedetomidine on Postoperative Delirium in Patients Undergoing Awake Craniotomies: a Randomized Controlled Trial
Brief Title: Effect of Dexmedetomidine on Postoperative Delirium After Awake Craniotomies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-01-04
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Dexmedetomidine; Delirium; Awake Craniotomy
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Active Comparator): The DEX group patients will be received dexmedetomidine intraoperatively.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): The placebo group patients will be received 0.9% saline intraoperatively.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — The 200ug dexmedetomidine will be diluted into a 50ml syringe and administered with continuous infusion at a rate of 0.2 µg/kg/hour until the end of dural closure.
  Arms: DEX group
Drug: 0.9% saline — The 0.9% saline is administered with the same volume at the same speed as the other group.
  Arms: Placebo group

SUMMARY:
Postoperative delirium (POD) is a common complication, and the incidence of POD ranges from 10% to 60%. Previous studies suggested that frontal approach and tumor located at the temporal lobe were independent risk factors for POD after supratentorial tumor resections. Therefore, patients undergoing awake craniotomies are high-risk populations for POD. A lot of trials show that dexmedetomidine might help to reduce the incidence of delirium in patients undergoing non-cardiac surgery. However, the impact of dexmedetomidine (DEX) on POD for patients undergoing awake craniotomies remains unclear. The purpose of this study was to investigate the effect of DEX on POD in patients undergoing awake craniotomies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing selective awake craniotomies.
* Age ≥18 years.
* Obtain written informed consent.

Exclusion Criteria:

* 1.Preoperative moderate and severe cognitive impairment (Montreal Cognitive Assessment, MoCA< 18).
* 2.Preoperative psychotropic medication within one year.
* 3.BMI≤18 or ≥30 Kg/ m2
* 4.Pregnant or lactating women.
* 5.History of traumatic brain injury or neurosurgery.
* 6.Severe bradycardia (heart rate less than 40 beats per minute), sick sinus syndrome or second-to-third degree atrioventricular block.
* 7.Severe hepatic or renal dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium. | postoperative 5 day.
  postoperative delirium is assessed by the combination of the Richmond Anxiety Scale (RASS) and the Confusion assessment method for intensive care unit (CAM-ICU) or the 3-minute diagnostic interview for CAM (3D-CAM) as applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, MD,Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li M, Liu M, Cui Q, Zeng M, Li S, Zhang L, Peng Y. Effect of dexmedetomidine on postoperative delirium in patients undergoing awake craniotomies: study protocol of a randomized controlled trial. Trials. 2023 Sep 25;24(1):607. doi: 10.1186/s13063-023-07632-2. PMID 37743486